CLINICAL TRIAL: NCT04172870
Title: Evaluation of Demographic Variables, Clinical Parameters, Inflammatory Markers and Viruses in Periodontitis Patients With Coronary Artery Diseases
Brief Title: Evaluation of Inflammatory Markers and Periodontal Viruses on Periodontitis Patients With CAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and Director of PG studies, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB/2017/260; FLL/IRC/01/2017 (Other: Frontier Lifeline Hospital)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis; Coronary Artery Disease
Keywords: Ebstein Barr Virus; Cytomegalovirus; Herpes Simplex Virus; Pentraxins; Toll Like Receptors
MeSH Terms: conditions — Periodontitis; Coronary Artery Disease; Herpes Simplex | interventions — Cytogenetic Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Subgingival plaque sample, Atherosclerotic plaque samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group I: Healthy group ( No generalised periodontitis and no CAD)
  Interventions: Diagnostic Test: Molecular analysis
- Group II: Generalised periodontitis patients without CAD
  Interventions: Diagnostic Test: Molecular analysis
- Group III: CAD patients without generalised periodontitis
  Interventions: Diagnostic Test: Molecular analysis
- Group IV: Generalised periodontitis with CAD
  Interventions: Diagnostic Test: Molecular analysis

INTERVENTIONS:
Diagnostic Test: Molecular analysis — RT- PCR

SUMMARY:
To assess and compare the demographic variables, periodontal parameters, cardiac parameters and the expression of periodontal viruses (CMV, HSV and EBV) and inflammatory biomarkers(PTX-3, TLR-2 & TLR-4) in periodontally healthy and generalized periodontitis patients with and without coronary artery disease(CAD).

DETAILED DESCRIPTION:
A total of 240 subjects will be recruited based on the power of the study. The selected subjects will be divided into four groups based on the inclusion and exclusion criteria.

1. GROUP I: 60 healthy subjects ( No generalised periodontitis and no CAD)
2. GROUP II: 60 generalised periodontitis subjects without CAD
3. GROUP III: 60 CAD subjects without generalised periodontitis
4. GROUP IV: 60 subjects with Generalised periodontitis and CAD

Sub-gingival plaque samples will be collected from the subjects of all the four groups. Coronary artery plaque samples will be collected from the patients who were indicated for coronary artery bypass graft surgery (CABG) among group III and group IV.

The demographic variables , periodontal parameters , cardiac parameters , expression of periodontal viruses and inflammatory biomarkers will be measured in all four groups ,

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients with 30 to 65 years of age group
3. Both genders
4. Patients should have minimum of 10 natural teeth.
5. In case of group III and IV patients with coronary heart disease to be included.

Exclusion Criteria

1. Patients who had undergone periodontal therapy within the previous 6 months.
2. Type I and II Diabetes mellitus
3. Sarcoidosis patients.
4. Carcinoma patients.
5. Rheumatic arthritis patients.
6. Tuberculosis patients.
7. Immunosuppressive conditions.
8. Patients with other inflammatory diseases.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Indian Population
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal Virus and Inflammatory Markers expression in periodontitis patients with coronary artery disease | 2 years
  Expression of EBV, CMV, HSV, Pentraxins, TLR 2 and TLR 4 using PCR

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, PhD, Principal Investigator — MeenakshiAmmal Dental College & Hospital
Locations (1):
- MeenakshiAmmal Dental College and Hospital, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No
Perio-Continuum link could be shared through publications

REFERENCES:
- [Background] Gurses KM, Kocyigit D, Yalcin MU, Canpinar H, Oto MA, Ozer N, Tokgozoglu L, Guc D, Aytemir K. Enhanced Platelet Toll-like Receptor 2 and 4 Expression in Acute Coronary Syndrome and Stable Angina Pectoris. Am J Cardiol. 2015 Dec 1;116(11):1666-71. doi: 10.1016/j.amjcard.2015.08.048. Epub 2015 Sep 11. PMID 26455385
- [Background] Jenny NS, Arnold AM, Kuller LH, Tracy RP, Psaty BM. Associations of pentraxin 3 with cardiovascular disease and all-cause death: the Cardiovascular Health Study. Arterioscler Thromb Vasc Biol. 2009 Apr;29(4):594-9. doi: 10.1161/ATVBAHA.108.178947. Epub 2009 Jan 22. PMID 19164811
- [Background] Imbronito AV, Marcelino SL, Grande SR, Nunes FD, Romito GA. Detection of human cytomegalovirus and epstein-barr virus in coronary atherosclerotic tissue. Braz J Microbiol. 2010 Jul;41(3):563-6. doi: 10.1590/S1517-83822010000300004. Epub 2010 Sep 1. PMID 24031529